CLINICAL TRIAL: NCT03500432
Title: A Novel, Repeatable, and Effective Local Anesthesia Method for Transperineal Prostate biopsy-a Single Center Randomized Controlled Trial
Brief Title: A Study of a New Local Anesthesia Method for Transperineal Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Military Medical University (Other)
Responsible Party: Principal Investigator, yinghao Sun, Principal Investigator, Second Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: SP-FA2018001
Record Dates: First submitted 2018-03-21; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Prostate Biopsy; Local Anesthesia
Keywords: transperineal prostate biopsy; local anesthesia; prostate cancer diagnosis
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- periprostatic group (Active Comparator): local anesthesia of trnasperineal prostate biopsy with subcutaneous local anesthesia+periprostatic block
  Interventions: Procedure: local anesthesia of trnasperineal prostate biopsy
- PAT group (Active Comparator): local anesthesia of trnasperineal prostate biopsy with subcutaneous local anesthesia+periapical triangle (PAT) block
  Interventions: Procedure: local anesthesia of trnasperineal prostate biopsy
- TPA switch group (Experimental): local anesthesia of trnasperineal prostate biopsy with subcutaneous local anesthesia+TPA switch (transperineal prostate biopsy local anesthesia switch) block
  Interventions: Procedure: local anesthesia of trnasperineal prostate biopsy

INTERVENTIONS:
Procedure: local anesthesia of trnasperineal prostate biopsy — three different block site with lidocaine
  Other Names: lidocaine, long injection needles

SUMMARY:
In comparison with transrectal prostate biopsy, transperineal prostate biopsy has the advantage of better sampling from the anterior area, low risk of infection, and no rectal bleeding. The main problems associated with the transperineal method are pain control and additional general or spinal anesthesia. Three types of anesthesia have been reported for transperineal prostate biopsy: (1) spinal anesthesia; (2) general anesthesia; and (3) local anesthesia. From the viewpoint of patient selection (general anesthesia is contraindicated in some patients) and medical cost, local anesthesia is the most suitable choice for prostate biopsy. Periprostatic block is the standard method of local anesthesia for this procedure. However, periprostatic block is insufficient for transperineal prostate biopsy due to high pain sensitivity in this region. A number of new methods to eliminate pain have been reported, including (1) periapical triangle (PAT) block, (2) paraprostatic plus sexual nerve block, and (3) periprostatic block plus pudendal block.However, there is no anatomical basis for some of these methods, and there have been no randomized controlled trials to evaluate their effectiveness, and some methods are technically difficult to learn. In the previous perineal nerve autopsy, we found that there are two branches leading into the prostate and anterior lateral prostatic tissue, which is the main site of puncture pain. There is a fixed position where the two branches appear. Therefore, this anatomical position block may be a useful site for local anesthesia. We named this location the 'transperineal prostate biopsy local anesthesia switch' (abbreviated as TPA switch). In order to validate its effect, we organized this clinical trail.

DETAILED DESCRIPTION:
Ninety patients scheduled for prostate biopsy will include in this study. The clinical trial validation process will be as follows: (1) all patients are randomly divided into three groups (Figure 1): group 1, subcutaneous local anesthesia+periprostatic block; group 2, subcutaneous local anesthesia+periapical triangle (PAT) block; group 3, subcutaneous local anesthesia+TPA switch (transperineal prostate biopsy local anesthesia switch) block; VAS scores for each puncture and complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 1. ready to be performed transperineal prostate biopsy; 2. fully understand the protocol and aggree to undergo prostate biopsy with local anesthesia which might be elder methods or new experimental method.

Exclusion Criteria:

* 1.do not have the history of anaphylaxis or local anesthetic intoxation； 2. cardiac dysfunction or coagulation dysfunction; 3. Rectal disease which can not allowed to plug the ultrasound probe in; 4.do not fully understand our protocol; 5. do not aggree our protocol.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
highest VAS scores | ask patients in 2 minutes after prostate biopsy
  the highest VAS (visual analogue scale) scores during the procedure in one patient. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. VAS is the most common pain scale for quantification of endometriosis-related pain and skin graft donor site-related pain. In detail, it is a 10-point categorical scale pain measurement. The score ranges from 0 to 10, and the no pain is 0, and highest pain is 10.

SECONDARY OUTCOMES:
Complications | during the procedures and 1 days after the procedure
  Complications associated with local anesthesia. The complication include: bleeding, intoxation of local anesthetic and anaphylaxis of local anesthetic.
main VAS scores | ask patients in 2 minutes after prostate biopsy
  the main VAS (visual analogue scale) scores during the procedure in one patient. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. VAS is the most common pain scale for quantification of endometriosis-related pain and skin graft donor site-related pain. In detail, it is a 10-point categorical scale pain measurement. The score ranges from 0 to 10, and the no pain is 0, and highest pain is 10.
patients movement | during the transperineal prostate biopsy
  During the procedure if there is movement of the body which will affect the process of prostate biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Yinghao 2 Sun, professor, Study Chair — Second Military Medical University
Locations (1):
- Changhai Hospital,Second Military Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No